CLINICAL TRIAL: NCT02336841
Title: A Study of the Feasibility and Effectiveness of the Addition of Self Help And Recovery Guide for Eating Disorders (SHARED) to Treatment as Usual for Anorexia Nervosa
Brief Title: Self-Help And Recovery Guide in Eating Disorders
Acronym: SHARED
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: King's College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 159490
Record Dates: First submitted 2015-01-08; First posted 2015-01-13 (Estimated); Last update posted 2015-01-13 (Estimated); Status verified 2015-01

CONDITIONS: Anorexia Nervosa
Keywords: Guided Self-Help; Peer Mentoring; Anorexia Nervosa; Eating Disorders
MeSH Terms: conditions — Anorexia Nervosa; Feeding and Eating Disorders | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): Participants in this condition will receive the guided self-help intervention.
  Interventions: Other: Treatment as usual + Recovery MANTRA
- Control (Active Comparator): Participants in this condition will not receive the guided self-help intervention. They will receive treatment as usual and weekly feedback on their eating disorder symptoms for a period of 6 weeks.
  Interventions: Other: Treatment as usual + feedback

INTERVENTIONS:
Other: Treatment as usual + Recovery MANTRA — Participants in this group will receive the guided self-help intervention including video-clips, a workbook, and guidance from peer mentors, and treatment as usual.
  Arms: Intervention
Other: Treatment as usual + feedback — Participants in this group will receive treatment as usual and feedback on their eating disorder symptoms.
  Arms: Control

SUMMARY:
The aim of this study is to test a novel guided self-help intervention for patients with Anorexia Nervosa. The 6-week intervention includes the use of self-help materials (i.e. a workbook and short video-clips) and weekly guidance from a peer mentor (i.e. a person recovered from Anorexia Nervosa). Self-reports will be completed at baseline, end of 6 weeks, and 6- and 12 months follow-up. Participants interested in taking part will be randomly allocated to one of two groups.

DETAILED DESCRIPTION:
This trial investigates whether a guided self-care intervention (Recovery MANTRA) is a useful addition to treatment as usual (TAU) for individuals with anorexia nervosa (AN). Recovery MANTRA, a 6-week self-care intervention supplemented by peer mentorship, is a module extension of the Maudsley Model of Treatment for Adults with AN and targets the maintenance factors identified by the cognitive-interpersonal model of the illness.

Patients accessing outpatient services for AN are randomised to either TAU or TAU plus Recovery MANTRA. Outcomes variables include changes in body weight at the end of the intervention (primary) and changes in body weight and eating disorder symptoms at immediate and extended follow-ups (6-months and 12-months; secondary). Change is also assessed for the domains identified by the theoretical model, including, motivation, hope, confidence to change, positive mood, cognitive flexibility, therapeutic alliance and social adjustment. Feedback from peer mentors is gathered to understand the impact of providing guidance on their own well-being.

Results from this exploratory investigation will determine whether a larger clinical trial is justifiable and feasible for this affordable intervention which has potential for high reach and scalability.

ELIGIBILITY:
Inclusion Criteria:

- Referral to one of the participating specialist adult outpatient eating disorder clinics with a primary DSM-5 diagnosis of Anorexia Nervosa or OSFED (Other Specified Feeding or Eating Disorder) with a body mass index (BMI; kg/m2) of 18.5 or below. OSFED will be defined as having features of Anorexia but missing at least two of the four diagnostic criteria.

Exclusion Criteria:

* Insufficient knowledge of English
* Severe mental or physical illness needing treatment in its own right (e.g. psychosis or diabetes mellitus).

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2015-01; Primary Completion 2016-12 (Estimated); Study Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
Changes in body weight at the end of the intervention | 3 years

SECONDARY OUTCOMES:
Changes in eating disorder symptoms at the end of the intervention and follow-up | 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- King's College London, London, United Kingdom

REFERENCES:
- [Derived] Cardi V, Albano G, Salerno L, Lo Coco G, Ambwani S, Schmidt U, Macdonald P, Treasure J. The Feasibility of Using Guided Self-Help in Anorexia Nervosa: An Analysis of Drop-Out From the Study Protocol and Intervention Adherence. Front Psychol. 2020 Apr 16;11:707. doi: 10.3389/fpsyg.2020.00707. eCollection 2020. PMID 32373032
- [Derived] Ambwani S, Cardi V, Albano G, Cao L, Crosby RD, Macdonald P, Schmidt U, Treasure J. A multicenter audit of outpatient care for adult anorexia nervosa: Symptom trajectory, service use, and evidence in support of "early stage" versus "severe and enduring" classification. Int J Eat Disord. 2020 Aug;53(8):1337-1348. doi: 10.1002/eat.23246. Epub 2020 Feb 17. PMID 32064663
- [Derived] Cardi V, Ambwani S, Crosby R, Macdonald P, Todd G, Park J, Moss S, Schmidt U, Treasure J. Self-Help And Recovery guide for Eating Disorders (SHARED): study protocol for a randomized controlled trial. Trials. 2015 Apr 16;16:165. doi: 10.1186/s13063-015-0701-6. PMID 25885697